CLINICAL TRIAL: NCT02905617
Title: Post Market Clinical Experience Study of the Sientra 207 High-Strength Cohesive Plus (HSC+) Breast Implants in Primary and Revision Augmentation Participants
Brief Title: Post Market Clinical Experience Study of Sientra 207 Breast Implants
Status: Terminated | Type: Observational
Why Stopped: Low enrollment
Sponsor: Tiger Biosciences, LLC. (Industry)
Responsible Party: Sponsor
Other Study IDs: CP-1008
Record Dates: First submitted 2016-09-09; First posted 2016-09-19 (Estimated); Last update posted 2023-07-03 (Actual); Status verified 2023-04

CONDITIONS: Breast Augmentation; Breast Revision-Augmentation
Keywords: Breast Augmentation; Breast Revision-Augmentation

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Primary Augmentation: Subjects undergoing general breast enlargement receiving Sientra Style 207 Silicone Gel Breast Implant.
  Interventions: Device: Sientra 207 Silicone Gel Breast Implant
- Revision Augmentation: Subjects undergoing revision surgery with Sientra Style 207 Silicone Gel Breast Implant to revise or improve the result of a primary breast augmentation surgery.
  Interventions: Device: Sientra 207 Silicone Gel Breast Implant

INTERVENTIONS:
Device: Sientra 207 Silicone Gel Breast Implant — The Sientra 207 Silicone Gel Breast Implant is a textured, round device with high-strength cohesive plus (HSC+) silicone gel fill.

SUMMARY:
A 12-month study to evaluate the clinical experience with Sientra 207 Silicone Gel Breast Implants

DETAILED DESCRIPTION:
This study is designed to prospectively collect surgeon and participant satisfaction with the Sientra 207 implants in primary and revision augmentation participants over a 12-month time frame.

ELIGIBILITY:
Inclusion Criteria:

1. Is a candidate for primary or revision breast augmentation and is at least 22 years of age,
2. Agrees to Sientra study requirements and to comply with office follow-up visits at months 3, 6 and 12.

Exclusion Criteria:

1. Does not meet the Investigator's standard eligibility for breast augmentation or revision surgery
2. Surgeon is planning to use acellular dermal matrix (ADM) or surgical mesh and/or recommend postoperative massage.

Min Age: 22 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Women who receive Sientra Silicone 207 Gel Breast Implants for primary augmentation or revision augmentation
Sampling Method: Non-Probability Sample
Enrollment: 113 (Actual)
Dates: Start 2016-08 (Actual); Primary Completion 2020-07-15 (Actual); Study Completion 2020-07-15 (Actual)

PRIMARY OUTCOMES:
Investigator Overall Satisfaction Questionnaire | 3 months
  The primary outcome measure of the study is to obtain the Investigator Overall Satisfaction with the device using a 5-point scale where 1=definitely dissatisfied with the device to 5=definitely satisfied with the device.
Investigator Overall Satisfaction Questionnaire | 6 months
  The primary outcome measure of the study is to obtain the Investigator Overall Satisfaction with the device using a 5-point scale where 1=definitely dissatisfied with the device to 5=definitely satisfied with the device.
Investigator Overall Satisfaction Questionnaire | 12 months
  The primary outcome measure of the study is to obtain the Investigator Overall Satisfaction with the device using a 5-point scale where 1=definitely dissatisfied with the device to 5=definitely satisfied with the device.

CONTACTS AND LOCATIONS:
Overall Officials: Sientra, Inc., Study Director — Sponsor GmbH
Locations (1):
- Sientra, Inc., Santa Barbara, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Schwartz MR, Haws MJ, Phillips G. Results of the Postmarket Clinical Study of the Sientra 207 Highly Cohesive Gel Breast Implants in Primary and Revision Augmentation. Plast Reconstr Surg. 2018 Apr;141(4S Sientra Shaped and Round Cohesive Gel Implants):40S-48S. doi: 10.1097/PRS.0000000000004353. PMID 29595717